CLINICAL TRIAL: NCT02150148
Title: Vegetable Garden Feasibility Trial to Promote Function in Older Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CA182508; R21CA182508-01 (NIH)
Record Dates: First submitted 2014-05-24; First posted 2014-05-29 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2015-11

CONDITIONS: Cancer
Keywords: breast cancer; prostate cancer; colorectal cancer; small intestine cancer; thyroid cancer; Hodgkin lymphoma; non-Hodgkin lymphoma; endometrial cancer; kidney cancer; cervical cancer; diet; exercise; physical activity; garden
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Thyroid Neoplasms; Hodgkin Disease; Lymphoma, Non-Hodgkin; Endometrial Neoplasms; Kidney Neoplasms; Uterine Cervical Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mentored Gardening Intervention (Experimental): Participants in this arm will be provided with either a raised bed garden or 4 earthboxes, gardening supplies, and plants and seeds. A master gardener from the Cooperative Extension will mentor them over the course of a year to plant three gardens (spring, summer and fall).
  Interventions: Behavioral: Experimental: Mentored Gardening Intervention
- Wait-List (Other): Participants in this arm will be provided with the same gardening supplies as the other group, but will receive them one year after enrollment in the study. They also will receive instruction from a master gardener from the Cooperative Extension at this time as well.
  Interventions: Behavioral: Experimental: Mentored Gardening Intervention

INTERVENTIONS:
Behavioral: Experimental: Mentored Gardening Intervention — receives raised bed or earthboxes and gardening supplies and instruction on vegetable gardening

SUMMARY:
Cancer survivorship has been claimed a national priority, with a call to develop effective interventions that can prevent, delay, or mitigate the adverse effects and comorbidities in this high risk population. Strong evidence exists that a healthful diet and regular physical activity can prevent many chronic diseases and improve physical function. More research however is needed to develop interventions that can produce long-term adherence to healthful lifestyle behaviors. This pilot study is based on the hypothesis that vegetable gardening interventions will be feasible and result in improvements in diet and exercise behaviors as well as improvements in physical functioning and well-being.

DETAILED DESCRIPTION:
The proposed feasibility study relies on the extant infra-structure of the Alabama Cooperative Extension Master Gardener Program. A total of 46 older (≥65 years) cancer survivors recently diagnosed with a loco-regionally staged cancer with a good prognosis (i.e., ≥ 80% 5-year survival) and with 2 or more physical function limitations will be recruited from select rural and urban counties in Alabama and randomized to 1-of-2 study arms: 1) an intervention group that receives a 1-year mentored vegetable gardening intervention that pairs cancer survivors with certified Master Gardeners, or 2) a usual care control group that is observed during the year, but receives the gardening supplies at study completion. Aims of this study are to: 1) explore the feasibility and acceptability of a mentored vegetable gardening intervention by assessing accrual, retention, adherence, fidelity, and possible adverse events, 2) obtain means and precision estimates, and explore between-arm differences on pre-post changes in physical function and secondary endpoints (e.g., quality of life, fruit & vegetable intake, physical activity, etc.), and 3) to explore participant factors associated with program efficacy (e.g., gender, comorbidity).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with a loco-regionally staged cancer associated with an 60% or greater 5-year survival rate (localized and regional staged breast, Hodgkin lymphoma, prostate, ovary, endometrial, colorectal and thyroid cancers; localized cervix, kidney/renal pelvis, non-Hodgkin lymphoma, oral cavity/pharynx, small intestine, bladder and soft tissue cancers; and in situ bladder & breast cancer); and distant Hodgkin Lymphoma, and Testicular cancers.
* resides in select counties in Alabama;
* completed primary curative cancer treatments, i.e., surgery, chemotherapy or radiation therapy;
* at higher risk of functional decline (≥ 1 physical function (PF) limitations as defined by the SF36 PF subscale);
* currently eats less than 5 servings of fruits and vegetables/day;
* exercises less than 150 minutes/ week;
* speaks, reads and writes in English
* reside in a location that can accommodate 4 or more Earthboxes or 1-raised bed (4'x 8'), and that get at least 4 hours of sun a day with running water;
* willing to be randomized to either study arm and participate in the follow-up.

Exclusion Criteria

* history of lymphedema flares and axillary node dissection of 10 or more lymph nodes on one side of the body;
* not competent due to mental health or other very serious comorbid conditions (e.g., severe orthopedic conditions or scheduled for a hip or knee replacement with 6 months, paralysis, unstable angina or who have experienced a myocardial infarction, congestive heart failure or pulmonary conditions that require hospitalization or oxygen within 6 months, stroke, degenerative neurological conditions);
* currently taking pharmacologic doses of warfarin (does not include doses taken to maintain a port); or
* plants a vegetable garden at least annually

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
feasibility | baseline to 12 months
  attainment of accrual target of 46 eligible enrolled participants, retention of at least 80% of participants over the 12-month study period and the absence of any serious events attributable to the intervention

SECONDARY OUTCOMES:
physical function | baseline to 12 months
  assessed via the SF 36 physical function subscale and the senior fitness battery
diet quality | baseline to 12 months
  assessed via the Diet History Questionnaire
physical activity | baseline to 12 months
  assessed via the CHAMPS questionnaire with accelerometry confirmation
quality of life | baseline to 12 months
  assessed via the SF-36
biomarkers of successful aging | baseline to 12 months
  assessed via blood (serum) levels of IL-6, VCAM, d-dimer and telomerase and finger/toenail and saliva measures of cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Demark-Wahnefried, PhD, RD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Blair CK, Madan-Swain A, Locher JL, Desmond RA, de Los Santos J, Affuso O, Glover T, Smith K, Carley J, Lipsitz M, Sharma A, Krontiras H, Cantor A, Demark-Wahnefried W. Harvest for health gardening intervention feasibility study in cancer survivors. Acta Oncol. 2013 Aug;52(6):1110-8. doi: 10.3109/0284186X.2013.770165. Epub 2013 Feb 26. PMID 23438359
- [Derived] Cases MG, Blair CK, Hendricks PS, Smith K, Snyder S, Demark-Wahnefried W. Sustainability capacity of a vegetable gardening intervention for cancer survivors. BMC Public Health. 2022 Jun 22;22(1):1238. doi: 10.1186/s12889-022-13644-5. PMID 35733142
- [Derived] Demark-Wahnefried W, Cases MG, Cantor AB, Fruge AD, Smith KP, Locher J, Cohen HJ, Tsuruta Y, Daniel M, Kala R, De Los Santos JF. Pilot Randomized Controlled Trial of a Home Vegetable Gardening Intervention among Older Cancer Survivors Shows Feasibility, Satisfaction, and Promise in Improving Vegetable and Fruit Consumption, Reassurance of Worth, and the Trajectory of Central Adiposity. J Acad Nutr Diet. 2018 Apr;118(4):689-704. doi: 10.1016/j.jand.2017.11.001. Epub 2018 Jan 2. PMID 29305129